CLINICAL TRIAL: NCT01185119
Title: The Effect of Native GLP-1 on Glucose Metabolism in the CNS During Hyperglycemia in Healthy Young Men Assessed by PET
Brief Title: Effect of GLP-1 on Glucose Metabolism in CNS Assessed by PET
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Birgitte Brock, asso. prof., Aarhus University, Aarhus
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H80-CP-O015
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2011-03

CONDITIONS: Healthy
Keywords: glucose uptake and metabolism in brain
MeSH Terms: interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GLP-1 (Active Comparator): During hyperglycemic clamp and GLP-1 versus placebo infusion 10 men will be CNS-PET scanned
  Interventions: Drug: native glp-1 (7-36)
- placebo (Placebo Comparator): During hyperglycemic clamp and GLP-1 versus placebo infusion 10 men will be CNS-PET scanned
  Interventions: Drug: native glp-1 (7-36)

INTERVENTIONS:
Drug: native glp-1 (7-36) — During hyperglycemic clamp and GLP-1 versus placebo infusion 10 men will be CNS-PET scanned
  Other Names: glucagon like peptide-1 (7-36)

SUMMARY:
10 healthy men will be PET-scanned (CNS) twice in random order with infusions of placebo or Native GLP-1 during hyperglycemic clamp to uncover the metabolic effects of GLP-1 in perspectives of intervention of macrovascular late diabetic pathology such as stroke and AMI. Earlier studies have revealed tendencies towards steady glucose metabolism in the CNS despite fluctuations in blood sugar when infusing native GLP-1.

DETAILED DESCRIPTION:
Background Type 2 diabetes (T2D) is epidemically increasing throughout the world. T2D is frequently associated with multiple complications, where particularly the macrovascular complications in the form of myocardial infarction with its possible complication of death or heart failure, cerebral infarction and limb amputation are responsible for a vast increase in morbidity and mortality in this group of patients. Apart from the individual burden on the patient, T2D puts massive pressure on national health economies.

It is well established that blood glucose lowering drugs, antihypertensive as well as lipid lowering drugs all play a pivotal role in the treatment of the type 2 diabetic subjects. Regarding glycemia, there are frequently side effects with the 'classic' drugs such as hypoglycemia, weight gain, heart failure, and so forth. Another important caveat is that employing the anti-hyperglycemic drugs either as monotherapy or in combination does not lower blood glucose to the targets as defined by the ADA. In other words novel anti-diabetic drugs are urgently required. However, the incretin concept has recently been inaugurated in the pharmacological scenario.

Glucagon-like peptide-1-receptors (GLP-1R) are abundant on alpha- and beta-cells in the pancreas, but are also present in the heart and CNS, especially in hypothalamic and hippocampal regions. A wide range of extrapancreatic effects of GLP-1 have been observed such as slowed gastric emptying and satiety-stimulating effects through hypothalamic mechanisms. Recent studies have showed interesting results regarding protection of the heart during ischemia, and protection of the brain in the acute phases of stroke have been proposed. Over-all GLP-1 seems to display effects in heart, brain, vessels, kidneys, muscles and liver(7).

To our knowledge, our group has in a very recent study been the first, by sophisticated metabolic techniques, together with Positron Emission Tomography (PET), to demonstrate that GLP-1 per se reduces cerebral glucose transport in total cerebral grey matter as well as individual grey matter regions, thereby suggesting that GLP-1 may protect the brain by limiting intracerebral glucose fluctuation when plasma glucose is increased. In other words, GLP-1 regulates blood brain barrier (BBB) glucose transfer at normal glycemia and presumably also during hyperglycemia(19).

Glucagon-like-peptide-1 (GLP-1): T2D is characterized by several hormonal and metabolic abnormalities such as dysfunction of insulin secretion, glucagon excess, impaired Glucagon-like-peptide-1 (GLP-1) secretion, and insulin resistance.

GLP-1 is an incretin hormone with numerous documented effects on the glycemic response. It is one of the most potent insulinotropic agents known and is secreted from L-cells in the gut mucosa in response to food ingestion. Effects on the islet-cells are (I) Amplification of glucose dependent stimulation of insulin secretion (II) Inhibition of glucagon secretion. In animal and cellular studies GLP-1 stimulates β-cell neogenesis, growth and differentiation, and in vitro inhibition of β-cell apoptosis is observed. Thus GLP-1 is also a β-cell growth factor. For now, treatment with GLP-1 has seldom caused hypoglycaemia in type 2 diabetic patients.

Hypotheses Based on the findings in the above-mentioned study, we hypothesize that Native GLP-1 during hyperglycemia will protect the brain in healthy men from hyperglycemia by reducing blood-brain-barrier glucose transport and brain glucose metabolism.

Aim: With well established methodology, to compare the effect of native GLP-1 and placebo, respectively, on the consumption of glucose in the CNS assessed by uptake of 18-fluro-deoxy-glucose (FDG) monitored by PET-scan of healthy young men during hyperglycemic pituitary-pancreatic clamp in the perspective of future prevention of macrovascular complications of diabetes and possibly other diseases such as Alzheimer's disease and other neurodegenerative and cardiac diseases.

The primary endpoint of the project: steady glucose metabolism in the brain during hyperglycemia with native GLP-1 infusion compared to placebo.

Design: Randomized, double-blinded crossover design. Every participant will be CNS-PET-scanned twice in random order with GLP-1 and placebo-infusions interrupted by a 3-4 week wash-out period between study days.

The study will be performed similarly to our previously conducted FDG/PET-study(21) and pancreatic clamp as done by Nielsen et al.(22)

Methods

GLP-1 is a natural peptide hormone that is degraded by the enzyme DPPIV after few minutes in the circulation. The remaining hormones utilized in this study, are used as tools in the investigational design and will not be used as medical compounds themselves.

Hormone doses

* Somatostatin (Ferring) 300 μg/hour(22)
* Insulin Actrapid (NOVO Nordisk) 0,12 mU/kg/minute (22)
* Glucagon (NOVO Nordisk, Glucagen) 0.6 ng/kg/minute(22)
* Growth hormone (NOVO Nordisk) 2 ng/kg/minute(22)
* Native GLP-1 (PolyPeoptide) 1,2 pmol/kg/minute (23) Pancreatic and hyperglycemic clamp Somatostatin is administered to inhibit endogenous production of GLP-1, insulin, glucagon, and growth hormone. Insulin, glucagon, and growth hormone are administered to achieve basal hormone levels. 20% glucose is infused to achieve hyperglycemic clamp with plasma glucose at 9 mM which is by experience the highest level of hyperglycemia possible while still avoiding breakthrough of natural counterregulatory hormones.

Ethics: Apart from its documented effect on glycemic control, GLP-1 has potential protective impact in the brain. Patients with type-2 diabetes carry a significantly increased risk of ischemic heart disease and stroke that has not been substantially reduced by current treatments. Preliminary data suggest that clinical use of GLP-1 can lead to improved prophylaxis against late diabetic complications, which can be achieved in this patient group in addition to improved glycemic control. This project is conducted to map the physiology of GLP-1 in heathy during hyperglycemia.

We believe the current study will provide deeper insight into the extra-pancreatic effects of GLP-1, with the particular aim to develop efficient prophylaxis against late diabetic cerebrovascular and cardiovascular complications, which outweighs the known adverse effects of the elements of the study.

The study will be conducted in accordance with the principles described in the Helsinki Declaration II and will not be initiated before acceptance is granted from the local Ethics Committee.

Written consent from participants is required before studies can be commenced, and all participants are covered by insurance according to "Bekendtgørelse af lov om patientforsikring" and "Lov om erstatning for lægemiddelskader".

Informed consent All participants will receive written and oral information about the purpose and the expected scientific value of the project as well as detailed description of all procedures and risks involved. Specifically, the participant will be told that participation is completely voluntary, and withdrawal is accepted at any stage during the investigation.

The project coordinator, Dr. Michael Gejl Jensen, will provide oral information and hand out written material including the general information brochure "Before you decide….." ("Før du beslutter dig…"). The participant is allowed an accompanying person for the duration of the meeting.

Written consent is collected after a minimum of 24 hours for further consideration. Both the responsible physician and the participant sign the consent, and the latter will be provided a copy.

Data management Source data (original documentation of clinical findings, printouts, lab results, and other details necessary to completely reconstruct each study) are stored in case report forms and a common database. All personal information is locked away and inaccessible to all but the investigators. Screening ID, randomization ID, and initials in the database identify participants. The initials will be erased from the database after completion of the study to ensure anonymity. A separate chart containing screening ID, randomization ID, initials, and personal data will be stored at another location to allow re-identification of source data. Social security numbers (Danish: CPR-numbers) are present on electronical charts, which are kept in the individual electronical patient charts on the hospital server. This information will only be accessible to personnel in the study-group and not to doctors treating the patients in any future hospitalization. Data will automatically be erased from the server after 15 years. The study will be disclosed to the local Data Monitoring Board.

Financial aspects Each participant will receive dkr 2400 as compensation.

The applicant will provide the needed work in accordance with present rules and contracts concerning research fellows at Institute of Pharmacology, University of Aarhus and the Research Unit, Department of Endocrinology (M), Aarhus University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed
* Caucasian
* Male
* Age > 20 years and < 50 years
* BMI 20-30 kg/m² -

Exclusion Criteria:

Diabetes og first degree relative diabetes

* Clinically significant liver- or kidney-disease (se-ALAT > 2 times upper reference, or se-Creatinin > 130 mM
* Anemia
* Other abnormal biochemical value
* Any of the following:

  * Heart disease
  * Liver disease
  * Kidney disease
  * Lung disease
  * Gastro-intestinal disease
  * Dyslipidemia (total serum-cholesterol > 8 mmol/l, total cholesterol/HDL cholesterol ratio > 8 or se-triglyceride > 3.5 mmol/l)
  * Endocrine disease (other than diabetes)
  * CNS disease
  * Hematological disease
  * Loss of more than 100 ml blood within the latest month of inclusion
  * Compliance problems
  * Abuse of alcohol or drugs
  * Smoking
  * Participation in a clinical research study within 3 months of inclusion
  * Allergy towards study hormones
  * Medication with any drugs with effects on the glucose-metabolism, including *glitazones

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
steady glucose metabolism in the brain during hyperglycemia with Native GLP-1 infusion compared to placebo. | june 2010 - dec 2010

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte Brock, asso.prof., Principal Investigator — University of Aarhus, Dept. of Pharmacology
Locations (1):
- Aarhus University, Institute of Pharmacology, Aarhus C, Aarhus, Denmark